CLINICAL TRIAL: NCT06662162
Title: Microcurrent Stimulation Therapy for Intermediate to Advanced Nonexudative Age-related Macular Degeneration (i-SIGHT2): a Multicentre, Randomised, Sham-controlled, Double-masked, Clinical Device Trial.
Brief Title: Microcurrent Stimulation Therapy for Intermediate to Advanced Nonexudative Age-related Macular Degeneration
Acronym: i-SIGHT2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: i-Lumen Scientific AUS PTY LTD (Industry)
Collaborators: i-Lumen Scientific, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ILS-AMD-202
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Age-Related Macular Degeneration; Age-related Macular Degeneration (ARMD); Intermediate AMD; Geographic Atrophy Secondary to Age-related Macular Degeneration
Keywords: AMD; Intermediate AMD; Dry AMD; Geographic Atrophy
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Intervention Model Description: 2:1 Randomization of active to sham therapy
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Active i-Lumen AMD therapy (Experimental): Active transpalpebral microcurrent therapy
  Interventions: Device: i-Lumen AMD
- Sham i-Lumen AMD therapy (Sham Comparator): Sham transpalpebral microcurrent therapy
  Interventions: Device: i-Lumen AMD

INTERVENTIONS:
Device: i-Lumen AMD — i-Lumen AMD transpalpebral microcurrent stimulation system

SUMMARY:
The goal of this clinical trial is to characterize the safety and effectiveness of the i-Lumen AMD transpalpebral microcurrent device and therapy in patients with intermediate to advanced nonexudative AMD.

Participants will:

* Undergo an initial loading regimen, followed by 7 maintenance over the course of 11 months.
* Participants will return monthly through Month 14 (3 months post-last treatment) for evaluation and monitoring.

ELIGIBILITY:
Key Inclusion Criteria:

* Presence of at least one large druse >125 microns in diameter due to AMD.
* BCVA letter score of 35 to 70 letters (inclusive) (Snellen equivalent 6/12 to 6/60 [20/40 to 20/200])

Key Exclusion Criteria:

* Any implanted electrical device(s) including deep brain stimulator, hearing or visual implants (i.e., cochlear implant, auditory brainstem implant, retinal prostheses), and/or cardiac defibrillator/pacemaker.
* Implanted metallic device within 20 cm of the Treatment electrode (study eye(s)) and/or the grounding electrode (base of the hairline on the back of the neck).
* Uncontrolled diabetes, defined as glycated haemoglobin (HbA1c) >10% (13.3 mmol/L).
* Current tobacco or tobacco-related product use or history within the past 5 years of heavy smoking (defined as, on average, more than half a pack of cigarettes per day).
* Known severe allergy to fluorescein dye.
* Medical diagnosis of severe dry eye defined as requiring either artificial tears more than six (6) times a day or prescription drops (i.e., Restasis, Xiidra, or Cequa).
* History of seizure disorders, chronic migraines and/or cluster headaches.
* History and/or evidence of diabetic retinopathy in either eye as assessed by CF, fundus fluorescein angiography (FA), and OCT, to be confirmed by the Central Reading Centre.
* Other conditions which pre-dispose to chorioretinal atrophy such as inherited retinal dystrophy (i.e., Stargardt's disease, Best's disease, pattern dystrophy, central areolar choroidal dystrophy, etc.).
* History and/or evidence of exudative AMD in the study eye as assessed by CF, FA (or OCT-A ), and OCT, to be confirmed by Central Reading Centre.
* GA involving the foveal centre, as assessed by the Central Reading Centre using AF and OCT.
* History of intravitreal injections for GA (e.g., Syfovre or Izervay).
* Treatment with photobiomodulation (PBM) therapy or short pulse laser within 12 months prior to screening.
* Glaucoma requiring ≥3 medications and/or drops per day, or history of trabeculectomy.
* History of any kind of intraocular surgery, excluding cataract surgery performed ≥3 months from Screening.
* History of yttrium aluminium garnet (YAG) laser posterior capsulotomy <1 month from Screening.
* Visually significant cataracts and/or visually significant posterior capsular opacification.
* History of amblyopia.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean Change BCVA from Baseline | Month 3
  Mean change in per-eye (treated study eye [unilateral] or treated primary study eye [bilateral]) from Baseline in distance BCVA letter score on the ETDRS VA chart, active vs sham.

SECONDARY OUTCOMES:
Portion of per-eye Responders | Month 3
  1. Difference in proportion of per-eye (treated study eye [unilateral] or treated primary study eye [bilateral]) gaining ≥10 letters from Baseline in distance BCVA ETDRS, active vs sham.
Mean Change BCVA from Baseline | Month 6
  Mean change in per-eye (treated study eye [unilateral] or treated primary study eye [bilateral]) from Baseline in distance BCVA letter score on the ETDRS VA chart, active vs sham.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Mundy, Study Director — i-Lumen Scientific AUS PTY LTD
Locations (9):
- Australia (5):
  - Eye Clinic Albury-Wodonga, Albury, New South Wales
  - Sydney Eye Hospital, Sydney, New South Wales
  - Hobart Eye Surgeons, Hobart, Tasmania
  - Adelaide Eye & Retina Centre, Adelaide, Victoria
  - Cerulea, East Melbourne, Victoria
- New Zealand (2):
  - Auckland Eye Limited, Remuera, Auckland
  - Southern Eye Specialist, Christchurch
- United Kingdom (2):
  - King's College Hospital, London
  - London North West University Healthcare, Middlesex

IPD SHARING:
Plan to Share IPD: No